CLINICAL TRIAL: NCT03980977
Title: Collection of Biological Samples for Stydy of Unusual Toxicity Induced by Radiotherapy
Brief Title: Unusual Toxicity Induced by Radiotherapy
Acronym: CRYOTOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017 A00266-47
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: unusual toxicity; radiosensitivity; radiotherapy; fibroblast cell; indirect immunofluorescence test
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skin and/or tumor Biopsy and blood sample (Other)
  Interventions: Other: skin biopsy; Other: tumor biopsy; Other: blood sample

INTERVENTIONS:
Other: skin biopsy — skin biopsy will be taken under local anesthesia using a patch of lidocaine and prilocaine. In practice, during the skin biopsy, the skin must be cleaned with chlorhexidine or alcohol, to the exclusion of any other antiseptic. The biopsy will preferably be done with a dermatome (or "punch", 12 G).
Other: tumor biopsy — an additional tumor sample will be taken during programmed diagnostic procedure.
Other: blood sample — blood sample will be taken for biological collection

SUMMARY:
In order to evaluate the physiopathological knowledge of the different pathological manifestations associated with individual radiosensitivity, it seems essential to carry out this pilot study. It has agglomerated homogeneous tissue samples to identify new biomarkers for patient diagnosis and follow-up, and may predict the therapeutic response. These knowledge will help to treatment customization.

ELIGIBILITY:
Inclusion Criteria:

* Child or teenager aged 2 to <18
* Man, Woman> 18 years old
* Patient with one of these situations:

  * Unusual toxicity in progress or after radiotherapy
  * Indication of radiotherapy and suspicion of abnormal pathways of response to ionizing radiation - constitutional (genetic disease) or acquired (systemic disease) - which may generate unusual radioinduced toxicity
* Patient information and informed consent signed by the patient. For children and teenager : information to parents and obtaining informed consent
* Affiliation to a social security scheme.

Exclusion Criteria:

* Contraindication for skin and / or tumoral biopsy
* Contraindication for blood sample of 2.5 ml
* Persons deprived of liberty or under supervision

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
skin fibroblast radiosensitivity | 2 to 3 months after skin biopsy
  The number of residual double strand break at 24 hours (number of 53BP1 foci) after a dose of 2 Gy will be quantified with indirect immunofluorescence

SECONDARY OUTCOMES:
tumor cells radiosensitivity | 2 to 3 months after tumor biopsy
  The number of residual double strand break at 24 hours (number of 53BP1 foci) after a dose of 2 Gy will be quantified with indirect immunofluorescence

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No